CLINICAL TRIAL: NCT02496481
Title: A Brief Motivational Interviewing Intervention in the Emergency Department to Increase Size-Appropriate Child Passenger Restraint Use
Brief Title: A Brief MI Intervention in the ED to Increase Child Passenger Restraint Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Hurley Medical Center (Other)
Responsible Party: Principal Investigator, Michelle L. Macy, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00096047
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Child Restraint Systems; Seat Belts
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group1 Baseline+MI+tailored brochure (Experimental): Participants randomized to Group 1 will receive the motivational interviewing intervention in the ED and will be mailed a tailored educational brochure about child passenger safety.
  All participants will complete the baseline assessment survey, a 2 week follow-up phone call and a 6 month follow-up encounter.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Tailored brochure
- Group2 Baseline+MI+general info (Experimental): Participants randomized to Group 2 will receive the motivational interviewing intervention in the ED and will be mailed a generic educational brochure about child passenger safety.
  All participants will complete the baseline assessment survey, a 2 week follow-up phone call and a 6 month follow-up encounter.
  Interventions: Behavioral: Motivational Interviewing
- Group3 Baseline+tailored brochure (Experimental): Participants randomized to Group 3 will receive no intervention in the ED and will be mailed a tailored educational brochure about child passenger safety
  All participants will complete the baseline assessment survey, a 2 week follow-up phone call and a 6 month follow-up encounter.
  Interventions: Behavioral: Tailored brochure
- Group4 Baseline+general info (No Intervention): Control Group. Participants randomized to this arm will receive no intervention in the ED and will be mailed a generic educational brochure about child passenger safety.
  All participants will complete the baseline assessment survey, a 2 week follow-up phone call and a 6 month follow-up encounter.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational interviewing (MI) in the ED has been used to encourage a variety of health behaviors among at-risk patients. In this study, researchers will employ motivational interviewing with half of the study participants to investigate the effects of the technique on child passenger restraint behaviors in a population of parents of children birth to 10 years of age.
  Arms: Group1 Baseline+MI+tailored brochure; Group2 Baseline+MI+general info
Behavioral: Tailored brochure — Tailored Print materials will be mailed to half of participants to investigate the effects of using patient-centered educational materials compared with generic educational materials to influence child passenger restraint behaviors in a population of parents of children birth to 10 years of age.
  Arms: Group1 Baseline+MI+tailored brochure; Group3 Baseline+tailored brochure

SUMMARY:
This study involves an emergency department (ED)-based intervention utilizing Motivational Interviewing (MI) techniques and patient-centered (e.g., tailored) print materials to promote the correct and consistent use of size-appropriate child passenger restraints (car seats, booster seats, and seat belts). This study is designed as a randomized pilot trial.

DETAILED DESCRIPTION:
Motor vehicle collisions (MVCs) remain a leading cause of death among children after the first year of life despite substantial improvements in passenger safety. Deaths and severe injuries from MVCs can be reduced significantly through the consistent use of size-appropriate child passenger restraints. Still, 10% of children ride completely unrestrained and roughly one-quarter do not use the recommended restraint for their size. New approaches are needed to motivate behavior change among parents who do not consistently use size-appropriate passenger restraints for their children from birth through age 10. Emergency department (ED) visits represent unique opportunities to reach vulnerable children and their parents who have difficulty accessing the primary care settings where childhood injury prevention information is commonly provided. Motivational interviewing (MI) in the ED has been used to encourage a variety of health behaviors among at-risk patients. However, MI has not been previously evaluated for child passenger safety promotion programs. This study will involve an ED-based intervention utilizing MI techniques and patient-centered (e.g., tailored) print materials to promote the correct and consistent use of size-appropriate child passenger restraints. This study is designed as a randomized pilot trial of the intervention utilizing a 2x2 factorial design to examine the independent and additive effects of ED-based MI and tailored print materials on the consistent use of size-appropriate child passenger restraints. Aim 1) To assess the feasibility and acceptability of the ED-based intervention among parents of children from birth through age 10; Aim 2) To determine the impact of the intervention on child passenger restraint attitudes and practices at 6-month follow-up in comparison to baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult (18+ years) parent or caregiver who regularly drives with their child,
* are able to speak and read English,
* who is presenting to the ED with their child age birth to 10 years.
* Child must be <4'9" in height.

Exclusion Criteria:

* Adult participants must be able to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Use of size-appropriate restraint | 6 month follow up
  At the 6-month follow-up encounter, we will reassess the child's current passenger restraint use. We will measure the impact of the intervention on use of a size-appropriate restraint for the child.

SECONDARY OUTCOMES:
Transition at the recommended time | 6 month follow up
  At the 6-month follow-up encounter, we will measure the impact of the intervention on the appropriateness of the transition to the next restraint.
Change in sub-optimal restraint use | 6 month follow up
  We will determine change from baseline to 6-month follow-up in parent's report of allowing sub-optimal restraint use (e.g., unrestrained, premature transition to a less protective restraint).
Acceptability of the intervention (composite measure) | 2 week follow up
  Participants will be asked to provide impressions of acceptability of the intervention by rating the following:
  * quality of educational information received in relation to the study
  * amount of time spent reviewing study educational materials
  * amount of information shared with family/friends
  * acceptability of initiating the intervention in the ED
Acceptability of the intervention (composite measure) | 6 month follow up
  Participants will be asked to provide impressions of acceptability of the intervention by rating the following:
  * quality of educational information received in relation to the study
  * amount of time spent reviewing study educational materials
  * amount of information shared with family/friends
  * acceptability of initiating the intervention in the ED

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan C.S. Mott Children's Hospital Emergency Department, Ann Arbor, Michigan
  - Hurley Medical Center Emergency Department, Flint, Michigan

IPD SHARING:
Plan to Share IPD: Undecided